CLINICAL TRIAL: NCT00317772
Title: A Phase I/II Study of Weekly Topotecan and Gefitinib (Iressa) in Patients With Platinum-Resistant Ovarian, Peritoneal, of Fallopian Tube Cancer
Brief Title: Topotecan and Gefitinib (Iressa) for Ovarian, Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: AstraZeneca (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2003-0322
Record Dates: First submitted 2006-04-21; First posted 2006-04-25 (Estimated); Results first posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Ovarian Cancer; Peritoneal Neoplasms; Fallopian Tube Cancer
Keywords: Epithelial Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer; Epidermal Growth Factor; Platinum Hypersensitivity; Hycamtin; Gefitinib; Iressa; Topotecan; EGFR
MeSH Terms: conditions — Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Topotecan; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Topotecan + Gefitinib (Experimental): Phase I: Topotecan: 2.0, 3.0, or 4.0 mg/m^2 by vein Days 1, 8 and 15 of 28 day cycle.
  Gefitinib: 250 mg by mouth daily.
  Phase II: Topotecan starting dose: MTD from Phase I by vein Days 1, 8, and 15 of 28 day cycle.
  Gefitinib: 250 by mouth daily for 28 Days.
  Interventions: Drug: Topotecan; Drug: Gefitinib

INTERVENTIONS:
Drug: Topotecan — Phase I Starting Dose: 2 mg/m^2 by vein Weekly Over 30 Minutes on Days 1, 8, and 15.
  Phase II: MTD dose from Phase I by vein weekly on Days 1, 8, and 15.
Drug: Gefitinib — Phase I: 250 mg by mouth daily for 28 Days.
  Phase II: 250 mg by mouth daily for 28 Days.
  Other Names: Iressa

SUMMARY:
The purposes of this study are:

1. To determine the dose limiting toxicity (DLT) and the maximum tolerated dose (MTD) weekly of topotecan in combination with standard dose gefitinib in patients with relapsed, platinum-resistant, ovarian, peritoneal or fallopian tube cancers that are epidermal growth factor receptor (EGF-R) positive (>/= 1+).
2. To determine the response rate and response duration in this patient population treated with the maximum tolerated dose (MTD) of topotecan administered on a weekly schedule in combination with standard dose gefitinib, given by way of the mouth (PO) daily.

DETAILED DESCRIPTION:
Gefitinib inhibits the activity of a molecule present on the cancer cell that plays a role in cancer cell growth. Topotecan is an FDA approved drug used to treat ovarian cancer that is still present after treatment with chemotherapy. It is also used to treat recurrent ovarian cancer (patients whose cancer returns after they have been cancer-free for a period of time).

Before treatment starts, you will have a complete physical exam, routine blood tests (about 2-3 teaspoons), a chest x-ray, and a CT scan or MRI. Women who are able to have children must have a negative blood pregnancy test.

There are 2 phases to this study. In the first phase, 3 different dose levels of topotecan are being studied. The dose of topotecan that you receive will depend on when you are enrolled. It will also depend on whether or not other participants had side effects from their treatment. Although the dose of topotecan will vary, the dose of gefitinib is the same for all participants. Up to 6 participants may be treated at each dose. The goal of this portion of the study is to find the highest safe dose of this drug combination. Up to 18 patients will be treated on this part of the study.

Once the highest safe dose of topotecan has been found, the second phase of the study will begin. In this phase, all participants will receive the same dose of topotecan and gefitinib. Up to 40 patients will be enrolled in this part of the study (but 6 will be from the 1st portion of the study.

Each treatment cycle is 28 days long. You will take one gefitinib tablet by mouth every day beginning on Day 1. In addition, you will be given topotecan through a catheter (tube) placed in a vein over 30 minutes on Days 1, 8, and 15.

Blood tests to check your kidney, liver, and bone marrow function and a complete checkup (physical examination, including a pelvic and rectal exam) will be done before each course of therapy and a month after treatment ends. About 2-3 teaspoons of blood will be collected for routine blood tests each time blood is drawn during this study. Follow up CT scans or MRI scans will be done after every 2 to 3 cycles to evaluate your response to treatment.

You will be taken off study if your disease gets worse or intolerable side effects occur. If you have a complete response to this therapy (no evidence of cancer) then treatment will continue for an additional 6 months and then stop. All treatment is given on an outpatient basis at UTMDACC.

You will be monitored for at least 30 days after your last dose of therapy. If you have side effects related to this treatment combination, you will be monitored longer (until the side effects have gone away).

This is an investigational study. Both gefitinib and topotecan are FDA approved and commercially available. However, their use together in this study is investigational. A total of up to 52 patients will take part in this study. All will be enrolled at UTMDACC.

ELIGIBILITY:
Inclusion Criteria:

* Women with platinum-resistant, histologically confirmed epithelial ovarian, fallopian tube or peritoneal cancer. Resistance is defined as: Progression of disease during platinum chemotherapy, or progression of disease within 6 months of completing platinum chemotherapy, or failure to achieve a complete response, with persistent macroscopic disease, after an adequate trial of primary therapy.
* EGF-R expression must be positive (e.g., 1+ or greater) See appendix G.
* Patients with a known hypersensitivity to platinum compounds, who have failed a desensitization regimen, or in the opinion of the investigator, are not good candidates for desensitization, are eligible.
* Patients must have measurable disease.
* Unlimited number of prior chemotherapy regimens are allowed.
* Zubrod performance status </= 2.
* Patients must have adequate hepatic, renal, and bone marrow function, defined as serum creatinine </= 2 mg/dl (estimated creatinine clearance 50 ml/min); total bilirubin < /=2.0 X the upper limit of normal (ULN); alanine aminotransferase (ALT) </= 2X ULN; white blood count (WBC) >/= 3,000/mm3; absolute neutrophil count (ANC) >/= 1,500/mm3; platelets >/= 100,000/mm3.
* At least three weeks must have elapsed from completion of chemotherapy or radiation therapy.
* At least 30 days must have elapsed from completion of treatment with a non-approved or investigational drug.
* Patients must sign an informed consent indicating that they are aware of the investigational nature of the study, in keeping with the policies of the hospital. The only approved consent is appended to this protocol.
* Women of childbearing potential must be willing to practice acceptable methods of birth control to prevent pregnancy.

Exclusion Criteria:

* Patients with borderline or low malignant potential tumors are not eligible.
* Patients who have had prior therapy with topoisomerase I inhibitors.
* Patients who are pregnant or lactating.
* Concurrent chemotherapy, radiation therapy, or surgery (excluding palliative radiation).
* Concurrent, uncontrolled, medical or psychiatric disorders.
* Patients with an active infection.
* Patients with a known hypersensitivity to topotecan or iressa.
* Patients with severe cardiovascular disease (i.e. arrhythmias requiring chronic treatment or congestive heart failure) (NYHA classification III or IV).
* History of other malignancy (except nonmelanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission and off all therapy for that disease for a minimum of 5 years.
* Patients with overt psychosis or mental disability or otherwise incompetent to give informed consent.
* Patients who have had prior anti-EGFR therapy (i.e. Tarceva, Cetuximab).
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the trial.
* Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St. John's Wort.
* Any evidence of clinically active interstitial lung disease (patient with chronic stable radiographic changes who are asymptomatic are eligible).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2004-09-02 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Levenback, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chelariu-Raicu A, Levenback CF, Slomovitz BM, Wolf J, Bodurka DC, Kavanagh JJ, Morrison C, Gershenson DM, Coleman RL. Phase Ib/II study of weekly topotecan and daily gefitinib in patients with platinum resistant ovarian, peritoneal, or fallopian tube cancer. Int J Gynecol Cancer. 2020 Nov;30(11):1768-1774. doi: 10.1136/ijgc-2020-001863. Epub 2020 Oct 9. PMID 33037105
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 09/02/2004 and closed to new patient entry on 01/10/2007. All recruitments were done in a medical clinic setting.
Groups:
- Phase 1 Dose Level 1: Topotecan 2 mg/m2 IV on Days 1, 8, and 15 plus daily Gefitinib 250 mg given PO
- Phase 1 Dose Level 2: Topotecan 3 mg/m2 IV on Days 1, 8, and 15 plus daily Gefitinib 250 mg given PO
- Phase 1 Dose Level 3; Expansion Phase: Topotecan 4 mg/m2 IV on Days 1, 8, and 15 plus daily Gefitinib 250 mg given PO
Period: Overall Study
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Expansion Phase
Started | 3 | 3 | 3 | 10
Completed | 1 | 1 | 2 | 1
Not Completed | 2 | 2 | 1 | 9
Not completed — Adverse Event | 0 | 0 | 0 | 2
Not completed — Disease Progression | 2 | 2 | 1 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Expansion Phase | Total
Number analyzed (Participants) | 3 | 3 | 3 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 1 | 7 | 13
  >=65 years | 0 | 1 | 2 | 3 | 6
Age, Continuous [Mean (Full Range); unit: years] | 55 [46 to 65] | 55 [42 to 76] | 68 [61 to 74] | 60 [47 to 71] | 60 [42 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 10 | 19
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 3 | 9 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1
  White | 3 | 3 | 3 | 7 | 16
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: Dose-limiting toxicity defined as any Grade 4 hematological toxicity and any > Grade 3 non-hematologic toxicity. The DLT (dose-limiting toxicity) is defined as any Grade 4 hematological toxicity and any > Grade 3 non-hematologic toxicity.
Time Frame: Continual reassessment method, prior to each 28 day cycle, an average of 60 days
Measure: Number; unit: Dose Limiting Toxicities
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3
Number analyzed (Participants) | 3 | 3 | 3
Dose Limiting Toxicities | 2 | 3 | 4

2. Primary Outcome: Maximum Tolerated Dose (MTD) of Topotecan
Description: Maximum tolerated dose is highest dose level in which 6 patients treated with at most 1 experiencing DLT.
Time Frame: At end of first course, prior to each new course (28 day cycle). Continual reassessment method (CRM) during each course for toxicity, an average of 60 days
Measure: Number; unit: mg/m^2
Groups:
- All Phase 1 Participants: Topotecan 4 mg/m2 IV on Days 1, 8, and 15 plus daily Gefitinib 250 mg given PO
Arm/Group | All Phase 1 Participants
Number analyzed (Participants) | 9
mg/m^2 | 4

3. Secondary Outcome: Response Rate
Description: Measurable disease defined as at least one lesion that can be accurately measured in at least one dimension. Complete Response (CR): disappearance of all target and non-target lesions and no evidence of new lesions. Partial Response (PR): At least 30% decrease in sum of longest dimensions (LD) of all target measurable lesions. Increasing Disease: At least a 20% increase in sum of LD of target lesions taking as reference smallest sum LD or appearance of new lesions within 8 weeks of study entry. Progression on existing non-target lesions, other than pleural effusions without cytological proof of neoplastic origin. Death due to disease without prior objective documentation of progression. Global deterioration in health status attributable to disease requiring a change in therapy without objective evidence of progression.
Time Frame: 61 weeks
Population: Two patients received only one cycle of treatment and therefore were not evaluable for response to therapy.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Expansion Phase
Number analyzed (Participants) | 3 | 3 | 3 | 10
Participants
  Complete response | 0 | 0 | 0 | 0
  Partial response | 1 | 0 | 1 | 0
  Stable disease | 0 | 1 | 1 | 1
  Progressive disease | 2 | 2 | 1 | 7
  Not evaluable | 0 | 0 | 0 | 2

ADVERSE EVENTS:
Time Frame: adverse events were accessed from baseline to 30 days following the last dose of study medication received, up to 2 years
Arm/Group | Phase 1 Dose Level 1 | Phase 1 Dose Level 2 | Phase 1 Dose Level 3 | Expansion Phase
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/10
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 9/10
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 Dose Level 1 (N=3) | Phase 1 Dose Level 2 (N=3) | Phase 1 Dose Level 3 (N=3) | Expansion Phase (N=10)
Hemoglobin (Blood and lymphatic system disorders) | 2 | 3 | 3 | 9
Neutrophils (Blood and lymphatic system disorders) | 2 | 3 | 2 | 6
Platelets (Blood and lymphatic system disorders) | 0 | 1 | 2 | 4
Febrile neutropenia (Infections and infestations) | 1 | 0 | 0 | 2
Dehydration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 4
Hypokalemia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 2 | 9
Mucositis (Gastrointestinal disorders) | 1 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 3 | 2 | 1 | 9
Diarrhea (Gastrointestinal disorders) | 3 | 3 | 3 | 9
Nausea (Gastrointestinal disorders) | 2 | 1 | 2 | 6
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2 | 3
Anorexia (Gastrointestinal disorders) | 1 | 3 | 1 | 3
ALT increase (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
AST increase (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Blood bilirubin increase (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 6
Fatigue (General disorders) | 3 | 3 | 3 | 9
Mood alterations (Nervous system disorders) | 3 | 2 | 2 | 2
Neuropathy (Nervous system disorders) | 2 | 2 | 2 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2005-09-07): https://cdn.clinicaltrials.gov/large-docs/72/NCT00317772/Prot_SAP_000.pdf